CLINICAL TRIAL: NCT00405652
Title: Measurement of Patient Reported Gastrointestinal (GI) and Health-related Quality of Life (HRQL) Outcomes in Liver Transplant Recipients (MyLiver)
Brief Title: Measurement of Gastrointestinal (GI) and Health-related Quality of Life (HRQL) Outcomes in Liver Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080ADE09
Record Dates: First submitted 2006-11-27; First posted 2006-11-30 (Estimated); Results first posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-02

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation, mycophenolate, GI problems, Quality of Life
MeSH Terms: interventions — Mycophenolic Acid

ARMS (1):
- Enteric-coated Mycophenolate sodium (Experimental): Enteric-coated Mycophenolate sodium (EC-MPS), administered orally twice a day to achieve a dose equimolar to the dose of Mycophenolate mofetil (MMF) the patient was taking at the time of study entry up to a maximum dose of 1440 mg.
  Interventions: Drug: Enteric-coated Mycophenolate sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS) — experimental
  Other Names: myfortic

SUMMARY:
Treatment with the immunosuppressive drug mycophenolate mofetil (MMF) may result in gastrointestinal (GI) complications in some patients. This study will assess if a switch from MMF to enteric-coated mycophenolate sodium (EC-MPS) results in improved GI and/or health-related quality of life in liver transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* Received liver transplant at least 3 months prior to study enrollment.
* Receiving immunosuppressive regimen that includes a calcineurin or mTOR inhibitor, and MMF at time of study enrolment. The patient must be stable on current immunosuppressive regimen. The MMF dose must be stable for at least 1 month prior to enrollment. Steroid use will be according to local practice.
* Patients can only be enrolled into the study if it is expected that treatment will continue at the same dose until study end (6-8 weeks after enrollment).
* Patients with a medical condition that necessitates MPA-treatment for probably the next 6- 8 weeks (time of study duration).
* Patients with at least mild overall Gastrointestinal (G)I complications as assessed by the GI complications Case Report Form(CRF).
* Eligible and willing to convert to Myfortic.
* At lease 18 years of age.
* Willing to provide written informed consent.
* Able to meet all study requirements including completing the questionnaires and completing 2 study visits.
* Patients receiving drugs that may cause GI symptoms such as bisphosphonates, minerals, vitamins, antibiotics or proton pump inhibitors (PPIs) have to be on a stable dose of these substances for at least 1 month prior to enrollment. Patients receiving these drugs can only be enrolled into the study, if it is expected that treatment will continue at the same dose until study end (6-8 weeks after enrollment).
* Females capable of becoming pregnant must have a negative pregnancy test within 7 days prior to or at baseline. Pregnancy test has to be repeated every 4 weeks. Females are required to practice an approved method of birth control for the duration of the study and for a period of 6 weeks following discontinuation of study medication, even where there has been a history of infertility.

Exclusion criteria:

* If applicable, GI symptoms assumed or know not to be caused by MPA therapy (e.g. oral bisphosphonates induced, infections diarrhea).
* Acute rejection <1 week prior to study enrollment
* Patients with Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) and or/ bilirubin values >=3 x Upper limit normal (ULN) (values available from the last routine assessment within 3 months are acceptable).
* Patients with serum creatinine values >=265 umol/L (values available from the last routine assessment within 3 month are acceptable).
* Patients with hemoglobin values <7g/dL and/or an absolute platelet count of <50 x 10^9/L and /or an absolute leukocytes count of <2.0 x10^9/L (values available from the last routine assessment within 3 month are acceptable.)
* Woman of child-bearing potential who is planning to become pregnant or is pregnant and/or lactating or who is unwilling to use effective means of contraception.
* Presence of psychiatric illness (i.e., schizophrenia, major depression) that, in the opinion of the site investigator, could interfere with study requirements.
* Undergoing acute medical intervention or hospitalization.
* Presence of a medical condition not related to a GI event at the time of visit, which requires immediate medical intervention.
* Any other medical condition that, in the opinion of the site investigator based on recall or chart review, interfere with completing the study, including but not limited to, visual problems or cognitive impairment.
* Receiving any investigational drug or have received any investigational drug within 30 days prior to study enrollment.
* Patients with hypersensitivity to mycophenolate sodium, mycophenolic acid, mycophenolic mofetil or other components of the formulation (e.g. lactose; see also SmPCs)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Nuremberg, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enteric-coated Mycophenolate Sodium
Started | 34
Completed | 30
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 34
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Changes in Gastrointestinal Symptom Severity and Health Related Quality of Life
Description: Change in Gastrointestinal symptom rating scale (GSRS) total score from baseline visit to follow-up visit 6-8 weeks after treatment. The GSRS has 5 subscales (reflux, diarrhea, constipation, abdominal pain, and indigestion) producing a mean subscale score ranging from 1 (no discomfort) to 7 (very severe discomfort). The GSRS total score was computed by the mean of the subscale scores.
Time Frame: Baseline, End of Study (6-8 weeks)
Population: Intent to Treat Population (No last Observation Carried Forward). The number of participants completing the GSRS at Baseline = 31 and at the End of Study= 29.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 31
Scores on a Scale
  Baseline (Visit 1) n=31 | 2.88 (0.66)
  End of Study (Visit 2) n=29 | 2.10 (0.78)

2. Secondary Outcome: The Number of Participants With Subclinical Rejection as Evaluated by a Change in Liver Enzymes
Description: The number of participants with subclinical rejection episodes as defined by a steroid-sensitive, clinically relevant increase of AST, ALT, gamma-GT, AP or bilirubin (i.e., elevation of one or more of these enzymes that was considered clinically relevant and showed resolution upon treatment with a slight increase of steroid dosage).
Time Frame: 12-20 weeks
Population: Intent to Treat
Measure: Number; unit: Participants
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 34
Participants | 6

ADVERSE EVENTS:
Arm/Group | Enteric-coated Mycophenolate Sodium
Serious Adverse Events (participants affected / at risk) | 4/34
Other Adverse Events (participants affected / at risk) | 23/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-coated Mycophenolate Sodium (N=34)
Faecaloma (Gastrointestinal disorders) | 1
Hepatitis c (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Transplant failure (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Glutamate dehydrogenase increased (Investigations) | 1
Alcoholism (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-coated Mycophenolate Sodium (N=34)
Abdominal distension (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 2
Feeling cold (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 3
Headache (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.